CLINICAL TRIAL: NCT03900650
Title: Men's Sexual Risk Behaviors: Alcohol, Sexual Aggression, and Emotional Factors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); Georgia State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: STUDY00008097; 5R37AA025212 (NIH)
Record Dates: First submitted 2019-03-28; First posted 2019-04-03 (Actual); Results first posted 2023-11-29 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Sexual Behavior; Alcohol Drinking; Sexual Aggression; Emotions
Keywords: Condom use resistance; Emotion dysregulation
MeSH Terms: conditions — Sexual Behavior; Alcohol Drinking | interventions — Alcoholic Beverages

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Alcoholic beverage, High Provocation Manipulation (Experimental): Participants will receive a dose of alcohol mixed in fruit juice designed to achieve a peak breath alcohol concentration of .08%. Participants then receive an experimental manipulation designed to evoke negative emotions such as frustration.
  Interventions: Behavioral: High provocation manipulation; Behavioral: Alcoholic beverage
- Non-alcoholic beverage, High Provocation Manipulation (Experimental): Participants will receive a beverage that does not contain alcohol (fruit juice only). Participants then receive an experimental manipulation designed to evoke negative emotions such as frustration.
  Interventions: Behavioral: High provocation manipulation; Behavioral: Non-alcoholic beverage
- Alcoholic beverage, Low provocation manipulation (Experimental): Participants will receive a dose of alcohol mixed in fruit juice designed to achieve a peak breath alcohol concentration of .08%. Participants receive an experimental manipulation designed to evoke positive emotions.
  Interventions: Behavioral: Low provocation manipulation; Behavioral: Alcoholic beverage
- Non-alcoholic beverage, Low provocation manipulation (Experimental): Participants will receive a beverage that does not contain alcohol (fruit juice only). Participants then receive an experimental manipulation designed to evoke positive emotions.
  Interventions: Behavioral: Low provocation manipulation; Behavioral: Non-alcoholic beverage

INTERVENTIONS:
Behavioral: High provocation manipulation — Participants will engage in a laboratory task and will then report their emotions following the task.
  Arms: Alcoholic beverage, High Provocation Manipulation; Non-alcoholic beverage, High Provocation Manipulation
Behavioral: Low provocation manipulation — Participants will engage in a laboratory task and will then report their emotions following the task.
  Arms: Alcoholic beverage, Low provocation manipulation; Non-alcoholic beverage, Low provocation manipulation
Behavioral: Alcoholic beverage — Participants will consume an alcoholic beverage (vodka mixed with fruit juice) that is the equivalent of 3-4 standard alcoholic drinks based on their body weight.
  Arms: Alcoholic beverage, High Provocation Manipulation; Alcoholic beverage, Low provocation manipulation
Behavioral: Non-alcoholic beverage — Participants will consume a nonalcoholic beverage (fruit juice) that is the isovolemic equivalent of 3-4 standard alcoholic drinks based on their body weight.
  Arms: Non-alcoholic beverage, High Provocation Manipulation; Non-alcoholic beverage, Low provocation manipulation

SUMMARY:
Although correct, consistent condom use can greatly reduce sexually transmitted infections and unplanned pregnancies, resistance of condom use is common among young adults. Young men's alcohol intoxication and sexual aggression history are predictive of greater condom use resistance and other sexual risk behaviors (e.g., unprotected sex). Moreover, emotional factors may play a role in these associations, suggesting a promising avenue for continued research. This project builds upon our prior research through investigation of the emotional mechanisms involved in young men's alcohol-related sexual risk behavior. This research addresses a critical knowledge gap and advances the field through the use of multiple methods designed to evaluate distal and proximal emotional factors implicated in alcohol-related sexual risk. Male drinkers aged 21-30 who use condoms inconsistently (N = 420) will first complete a screening procedure followed by a baseline survey that will assess relevant constructs, including emotional traits, emotion dysregulation tendencies, and alcohol expectancies. They will then complete a 30-day daily diary assessment of their daily emotional states, daily coping motives pertaining to drinking and sex, and daily drinking and sexual risk behaviors to evaluate daily relationships among these factors. The same participants will complete an in-lab experiment assessing in-the-moment effects of alcohol intoxication and provocation on emotional states and sexual risk intentions. Statistical analyses will be used to examine the daily influence of emotional states and coping motives on alcohol consumption and sexual risk behaviors and the experimental effects of alcohol intoxication and provocation on emotional states and other mediators, as well as sexual risk intentions. Moderating effects of emotion dysregulation tendencies will also be examined, and the linkages between event-level and experimental relationships will be investigated. This research is both significant and innovative in that it will address the public health concern of men's sexual risk behaviors, including condom use resistance; will evaluate the role of emotional processes in men's alcohol-related sexual risk; and will use multiple methods to gather complementary types of data that will elucidate the mechanisms underlying alcohol-related sexual risk behaviors and provide an empirical evidence base from which to develop and inform prevention and intervention programs.

ELIGIBILITY:
Inclusion Criteria:

* Single
* Male
* Ages 21-30
* Engagement in unprotected intercourse with a woman at least once in the past year -
* Consumed alcohol at least 2 times per week in the past 30 days
* Had sex with a woman at least 2 times in the past 30 days

Exclusion Criteria:

* A history of alcohol problems
* A medical condition and/or medications which contraindicate alcohol consumption
* In a relationship that is monogamous and has lasted longer than 6 months

Ages: 21 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Self-defined as male
Enrollment: 420 (Actual)
Dates: Start 2019-03-07 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2023-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Davis, PhD, Principal Investigator — Arizona State University
Locations (1):
- Arizona State University, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
We will make available individual, de-identified participant data that underlie disseminated results.
Supporting Information: SAP
Time Frame: Immediately following publication and ending 3 years following publication.
Access Criteria: Researchers who provide a methodologically sound proposal for the use of the data.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Prior to assignment to an arm, 420 participants were enrolled, then completed an in-lab baseline session. They then completed 32 days of daily surveys. Participants then returned to the lab for a second session where they were assigned to a study arm.
Period: Overall Study
Arm/Group | Alcoholic Beverage, High Provocation Manipulation | Non-alcoholic Beverage, High Provocation Manipulation | Alcoholic Beverage, Low Provocation Manipulation | Non-alcoholic Beverage, Low Provocation Manipulation
Started | 74 | 75 | 74 | 70
Completed | 72 | 74 | 74 | 70
Not Completed | 2 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0
Not completed — Withdrawn by staff | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alcoholic Beverage, High Provocation Manipulation | Non-alcoholic Beverage, High Provocation Manipulation | Alcoholic Beverage, Low Provocation Manipulation | Non-alcoholic Beverage, Low Provocation Manipulation | Total
Number analyzed (Participants) | 74 | 75 | 74 | 70 | 293
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.96 (74) | 24.45 (2.98) | 24.27 (2.76) | 24.53 (2.74) | 24.39 (2.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 74 | 75 | 74 | 70 | 293
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 18 | 6 | 15 | 59
  Not Hispanic or Latino | 53 | 56 | 67 | 55 | 231
  Unknown or Not Reported | 1 | 1 | 1 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1 | 2
  Asian | 4 | 3 | 3 | 2 | 12
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 0 | 0 | 2
  Black or African American | 2 | 2 | 2 | 4 | 10
  White | 52 | 54 | 58 | 53 | 217
  More than one race | 10 | 12 | 8 | 7 | 37
  Unknown or Not Reported | 3 | 4 | 3 | 3 | 13
Region of Enrollment [Number; unit: participants]
  United States | 74 | 75 | 74 | 70 | 293

OUTCOME MEASURES:

1. Primary Outcome: Mean Score of Sexual Risk Intentions
Description: Scale name: Intentions to have unprotected sex Construct: Self-reported ratings of unprotected sex likelihood in a hypothetical scenario Scale range: 1 (not at all likely) to 7 (very likely) A higher value is a worse outcome. This is one total scale (no subscales). Items are averaged to compute a mean score.
Time Frame: within one hour of receiving the intervention
Population: Of the 293 participants, 3 withdrew before completing this measure. 6 participants had missing data on this measure. Thus, the analysis population for this outcome was 284.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Alcoholic Beverage, High Provocation Manipulation | Non-alcoholic Beverage, High Provocation Manipulation | Alcoholic Beverage, Low Provocation Manipulation | Non-alcoholic Beverage, Low Provocation Manipulation
Number analyzed (Participants) | 72 | 72 | 72 | 68
score on a scale | 2.35 (1.74) | 1.67 (1.26) | 2.15 (1.46) | 1.37 (.91)
Statistical Analysis 1: Comparison: Alcoholic Beverage, High Provocation Manipulation vs Non-alcoholic Beverage, High Provocation Manipulation vs Alcoholic Beverage, Low Provocation Manipulation vs Non-alcoholic Beverage, Low Provocation Manipulation; Test type: Other; p < .01, ANOVA; Mean Difference (Final Values) = 7.32

2. Primary Outcome: Sexual Risk Behavior
Description: Number of unprotected sexual intercourse events
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: Unprotected sex events
Arm/Group | Alcoholic Beverage, High Provocation Manipulation | Non-alcoholic Beverage, High Provocation Manipulation | Alcoholic Beverage, Low Provocation Manipulation | Non-alcoholic Beverage, Low Provocation Manipulation
Number analyzed (Participants) | 74 | 75 | 74 | 70
Unprotected sex events | 4.13 (4.32) | 3.34 (3.73) | 3.80 (4.65) | 3.69 (3.56)
Statistical Analysis 1: Comparison: Alcoholic Beverage, High Provocation Manipulation vs Non-alcoholic Beverage, High Provocation Manipulation vs Alcoholic Beverage, Low Provocation Manipulation vs Non-alcoholic Beverage, Low Provocation Manipulation; Test type: Other; p = .770, ANOVA — This p-value tests the effect of the study arms on number of sex events; Mean Difference (Final Values) = .377

ADVERSE EVENTS:
Time Frame: 6-8 weeks
Arm/Group | Alcoholic Beverage, High Provocation Manipulation | Non-alcoholic Beverage, High Provocation Manipulation | Alcoholic Beverage, Low Provocation Manipulation | Non-alcoholic Beverage, Low Provocation Manipulation
All-Cause Mortality (participants affected / at risk) | 0/74 | 0/75 | 0/74 | 0/70
Serious Adverse Events (participants affected / at risk) | 0/74 | 0/75 | 0/74 | 0/70
Other Adverse Events (participants affected / at risk) | 0/74 | 0/75 | 0/74 | 0/70

LIMITATIONS AND CAVEATS:
Data collection was paused for approximately 11 months due to COVID-19 safety protocols.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-18): https://cdn.clinicaltrials.gov/large-docs/50/NCT03900650/Prot_SAP_000.pdf